CLINICAL TRIAL: NCT03434145
Title: Changes of Ocular Structures After Hemodialysis in Patients With Chronic Kidney Diseases
Status: Completed | Type: Observational
Sponsor: Hanyang University (Other)
Responsible Party: Principal Investigator, Yong Un shin, Assistant professor, Hanyang University
Other Study IDs: 2016-05-005
Record Dates: First submitted 2018-02-05; First posted 2018-02-15 (Actual); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Chronic Kidney Diseases; Hemolysis
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hemolysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with chronic kidney diseases: patients with end stage retinal disease undergoing hemodialysis underwent various ophthalmologic exams before and after hemodialysis.
  Interventions: Other: ophthalmologic exams

INTERVENTIONS:
Other: ophthalmologic exams — ophthalmologic exams such as vision, intraocular pressure, axial length and optical coherence tomography

SUMMARY:
To evaluate the effect of hemodialysis on various ophthalmologic parameters in patients with end-stage kidney disease (ESRD).

DETAILED DESCRIPTION:
Subjects: patients with ESRD undergoing hemodialysis at the Dialysis Center of Hanyang Guri Hospital

Ocular parameters: visual acuity, intraocular pressure, axial length, OCT Other systemic parameters: body weight, ultrafiltration volume, and systolic/diastolic blood pressure

All measurements were performed near the dialysis center. Measurements were performed on Monday (for patients who underwent dialysis sessions on Monday, Wednesday, and Friday) or Tuesday (for patients who underwent dialysis sessions on Tuesday, Thursday, and Saturday.

All parameters were measured before and after the hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* 1) patients who are regularly dialyzed in our dialysis room to participate in the study
* 2) patients who agree with our study protocol
* 3) patients who have unstable general condition

Exclusion Criteria:

* 1) previous intraocular surgery, (2) baseline IOP greater than 22 mmHg, (3) presence of glaucomatous optic disc changes including excavation, thinning, or notching of the neuroretinal rim, (4) axial length greater than 26 mm, and (5) combined macular and retinal diseases such as central serous chorioretinopathy and age-related macular degeneration, except diabetic retinopathy.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with end-stage renal disease who undergoing hemodialysis
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-09-09 (Actual); Primary Completion 2017-09-07 (Actual); Study Completion 2017-12-29 (Actual)

PRIMARY OUTCOMES:
changes of retinal and choroidal thickness after hemodialysis | immediately (within 10 minutes) before and after hemodialysis
  retinal & choroidal thickness on OCT

SECONDARY OUTCOMES:
changes of foveal vascular density using optical coherence tomography-angiography (OCTA) after hemodialysis | immediately (within 10 minutes) before and after hemodialysis
  vessel density on OCTA
the effect of hemodialysis (HD) on anterior chamber angle by anterior segment optical coherence | immediately (within 10 minutes) before and after hemodialysis
  intraocular pressure, retinal thickness, anterior chamber angle

CONTACTS AND LOCATIONS:
Overall Officials: Heeyoon Cho, MD, Study Chair — Hanyang University

IPD SHARING:
Plan to Share IPD: No